CLINICAL TRIAL: NCT06860087
Title: Impact of Chromium Supplementation on Glucido-lipidic Metabolism, Oxidative Stress and Inflammatory State in Pregnant Women with Gestational Diabetes Mellitus
Brief Title: Impact of Chromium Supplementation on Glucido-lipidic Metabolism, Oxidative Stress and Inflammatory State in Patients with Gestational Diabetes
Acronym: Cr and GDM
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kasdi Merbah (Other)
Responsible Party: Principal Investigator, Hadjer SAIFI, Doctor of Biological Sciences, University Lecturer, Hopital Mouhamed Boudiaf, Ouergla, Algeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EA02/2025
Record Dates: First submitted 2025-02-15; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Gestational Diabetes Mellitus (GDM); Oxidative Stress; Inflammatory Status; Insulin Resistance; Leptin Resistance; Glucose Metabolism Disorder; Lipid Metabolism Disorders
Keywords: Inflammatory status markers; Oxidative stress markers; Glucido-lipidic metabolism; HOMA-IR; Leptin level; Lipid profile; Fasting plasma glucose; Insulin level
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance; Glucose Metabolism Disorders; Lipid Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: Our study will include 04 groups:
  1. Group of pregnant women with gestational diabetes supplemented with 200 µg/day of chromium picolinate
  2. Group of pregnant women with gestational diabetes supplemented with 400 µg/day of chromium picolinate
  3. Group of pregnant women with gestational diabetes not supplemented (diabetic control group)
  4. Group of healthy pregnant women not supplemented (healthy control group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Women with gestational diabetes mellitus supplemented with 200 µg/day of chromium picolinate (Active Comparator): 50 Pregnant women with gestational diabetes mellitus will receive an oral supplementation of 200 µg of chromium picolinate (Nutraxin, B'IOTA Laboratories, Istanbul, Turquie) per day for 06 weeks.
  Interventions: Dietary Supplement: Oral chromium supplementation during gestational diabetes mellitus through the administration of chromium picolinate tablets (200 µg/d)
- Women with gestational diabetes mellitus supplemented with 400 µg/day of chromium picolinate (Active Comparator): 50 Pregnant women with gestational diabetes mellitus will receive an oral supplementation of 400 µg of chromium picolinate (Nutraxin, B'IOTA Laboratories, Istanbul, Turquie) per day for 06 weeks.
  Interventions: Dietary Supplement: Dietary Supplement: Oral chromium supplementation during gestational diabetes mellitus through the administration of chromium picolinate tablets (400 µg/d)
- Pregnant women with gestational diabetes mellitus (Dibetic control group) (No Intervention): 50 pregnant women with gestational diabetes who will not take any supplements will undergo two fasting blood draws. One during the 28th week of pregnancy and the other at the end of the 34th week, to assess biomarkers of glucose and lipid metabolism, oxidative stress, and inflammation.
- Healthy pregnant women (Healthy control group) (No Intervention): 50 healthy pregnant women who will not take any supplements will undergo two fasting blood draws. one during the 28th week of pregnancy and the other at the end of the 34th week, to assess biomarkers of glucose and lipid metabolism, oxidative stress, and inflammation.

INTERVENTIONS:
Dietary Supplement: Oral chromium supplementation during gestational diabetes mellitus through the administration of chromium picolinate tablets (200 µg/d) — 50 Pregnant women with gestational diabetes mellitus will receive an oral supplementation of 200 µg of chromium picolinate (Nutraxin, B'IOTA Laboratories, Istanbul, Turquie) per day for 06 weeks, starting from their 28th week of pregnancy. 02 fasting blood samples will be taken: one just before the supplementation begins and the other upon its completion, to assess biomarkers of glucose and lipid metabolism, oxidative stress, and inflammation.
  Arms: Women with gestational diabetes mellitus supplemented with 200 µg/day of chromium picolinate
Dietary Supplement: Dietary Supplement: Oral chromium supplementation during gestational diabetes mellitus through the administration of chromium picolinate tablets (400 µg/d) — 50 Pregnant women with gestational diabetes mellitus will receive an oral supplementation of 400 µg of chromium picolinate (Nutraxin, B'IOTA Laboratories, Istanbul, Turquie) per day for 06 weeks, starting from their 28th week of pregnancy. 02 fasting blood samples will be taken: one just before the supplementation begins and the other upon its completion, to assess biomarkers of glucose and lipid metabolism, oxidative stress, and inflammation.
  Arms: Women with gestational diabetes mellitus supplemented with 400 µg/day of chromium picolinate

SUMMARY:
Our study aims to explore the influence of dietary chromium supplementation in the form of chromium picolinate, at different doses (200 µg and 400 µg per day), on the health of pregnant women with gestational diabetes. This study will also provide more information on the safety of this type of supplementation during pregnancies complicated by gestational diabetes mellitus.

The main questions it aims to answer are:

* Does chromium supplementation at various doses in women with gestational diabetes mellitus truly influence their glucido-lipidic metabolism, oxidative/antioxidant balance, and inflammatory state? If so, is it beneficial or detrimental?
* If this supplementation is beneficial, which dose is the most appropriate?
* Do these types of supplementation have any side effects on the health of the mother and fetus? The participants will take chromium supplements for 6 weeks (supplemented groups) while the control participants will not take them (healthy and diabetic control groups).

Chromium-supplemented participants will undergo a medical check-up every 02 weeks to closely monitor their health status and detect any potential side effects at an early stage.

Researchers will compare the biochemical profile, oxidative stress status, and inflammation markers between chromium-supplemented and non-supplemented participants to assess the impact of this trace element.

Researchers will compare the effects of chromium supplements at different doses with each other.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women:

  * Whose their gestational age is 28 weeks
  * They have no pathology or complication associated with their pregnancy.
* Pregnant women with gestational diabetes mellitus:

  * They will be selected according to the criteria of the one-step method for screening for gestational diabetes mellitus established by the WHO.
  * They have no other pathology or complication associated with pregnancy.
  * They are subjected to insulin therapy and a low-calorie diet, rich in protein, fiber and beneficial lipids (they will all asked to keep their medical treatment prescribed by their doctor).
* All women involved in this study will be systematically supplemented with 60 mg/d iron and 400 mg/d vitamin B9 during pregnancy as recommended by WHO.

Exclusion Criteria:

* Pregnant women with unrecognized diabetes, type I or type II, will not be involved in this study.
* Pregnant women who were supplemented before one month or during pregnancy, or who will need other micronutrient supplements during the study to avoid their influence on the results.
* Pregnant women who develop other health complications will be removed from the study and replaced by others.
* Women with gestational diabetes mellitus who were unable to complete chromium supplementation up to 6 weeks will be excluded from the study and replaced by others.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant biological women
Enrollment: 200 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Plasma chromium level (ng/dL) | At baseline and after six weeks
  In all groups by using Atomic Absorption Spectroscopy.
Fasting plasma glucose level (g/L) | At baseline and after six weeks
  In all groups, by a spectrophotometric method using a commercial kit.
Plasma cholesterol level (g/L) | At baseline and after six weeks
  In all groups, by spectrophotometric method using commercial kit.
Plasma triglyceride level (g/L) | At baseline and after six weeks
  In all groups, by spectrophotometric method using commercial kit.
Plasma total antioxidant status (mmol/L) | At baseline and after six weeks
  In all groups, by a spectrophotometric method using a commercial kit.
Erythrocyte glutathione peroxidase (U/g Hb) | At baseline and after six weeks
  In all groups, by a spectrophotometric method using a commercial kit.
Erythrocyte catalase (U/g Hb) | At baseline and after six weeks
  In all groups, by a spectrophotometric method using a commercial kit.
Erythrocyte superoxide dismutase (U/g Hb) | At baseline and after six weeks
  In all groups, by a spectrophotometric method using a commercial kit.
Plasma 8-Hydroxydeoxyguanosine (ng/mL) | At baseline and after six weeks
  In all groups, by spectrophotometric method using commercial kit.
Erythrocye malondialdehyde (µm/L) | At baseline and after six weeks
  In all groups, by spectrophotometric method using commercial kit.
Erythrocyte carbonyl protein (µm/L) | At baseline and after six weeks
  In all groups, by spectrophotometric method using commercial kit.
Plasma tumor necrosis factor-α (pg/mL) | At baseline and after six weeks
  In all groups, by spectrophotometric method using commercial kit.
Plasma interleukin-10 (pg/mL) | At baseline and after six weeks
  In all groups, by spectrophotometric method using commercial kit.
Plasma insulin level (µU/mL) | At baseline and after six weeks
  In all groups, by immunological method using commercial kit.

SECONDARY OUTCOMES:
Plasma leptin level (ng/mL) | At baseline and after six weeks
  In all groups, by an immunoenzymatic method using a commercial kit.
Age (year) | At baseline
Body Weight (kg) | At baseline and after six weeks
  Using an electronic balance
Height (m) | At baseline
Body Mass Index (kg/m^2) | At baseline and after six weeks
  Body mass index is a numerical value calculated using body weight (kg) and height (m) to determine whether they are suitable.
Plasma urea (g/L) | At baseline and after six weeks
  In all groups, by a spectrophotometric method using a commercial kit.
Plasma creatinine (mg/L) levels | At baseline and after six weeks
  In all groups, by a spectrophotometric method using a commercial kit.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Boudiaf Hospital, Ouargla, Ouargla, Ouargla Province, Algeria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP